CLINICAL TRIAL: NCT04204330
Title: Federal Cardiomonitoring System. Determination of the Efficiency of a Single-lead ECG Recorded with CardioQVARK Cardiac Monitor in Order to Detect Atrial Fibrillation in Primary Health Centers.
Brief Title: Federal Cardiomonitoring System. Determination of the Efficiency of a Single-lead ECG Monitor.
Acronym: FECAS-AFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 081018
Record Dates: First submitted 2019-12-07; First posted 2019-12-18 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; electronic health; mobile health
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CardioQVARK group (Experimental): Inclusion criteria:
  1. Males and females aged 20 to 96 years having one or more of the following risk factors:
     * hypertensive heart disease;
     * history of ischemic stroke or transient ischemic attacks;
     * type 1 and 2 diabetes;
     * class 1-3 obesity;
     * heart failure or decreased tolerance to physical activity due to dyspnea;
     * coronary artery disease (CAD) or chest pain without established CAD diagnosis;
     * peripheral artery atherosclerosis;
     * abnormal heart rhythms (episodes of palpitations, pauses in heartbeat).
  2. A patient's consent to participate in the study and the ability to sign an informed consent form.
  Exclusion criteria:
  1. acute coronary syndrome;
  2. acute ischemic or hemorrhagic stroke;
  3. mental illness;
  4. severe concomitant disease with life expectancy less than 2 years.
  Withdrawal criteria:
  1. Refusal to participate in the study.
  Interventions: Device: CardioQvark cardiac monitor and software, single-lead ECG

INTERVENTIONS:
Device: CardioQvark cardiac monitor and software, single-lead ECG — Registration certificate for the medical device No. РЗН 2019/8124 dated February 15, 2019.
  Product form: phone case.
  Way of applying:
  1. Download the CardioQVARK mobile application; create a profile.
  2. Fill out the questionnaire:
     * age;
     * date of birth;
     * sex;
     * weight;
     * height;
     * blood type;
     * eye color;
     * hair color;
     * occupation;
     * town;
     * alcohol consumption;
     * tobacco use;
     * overeating;
     * insufficient sleep;
     * hypertension;
     * type 2 diabetes;
     * pacemaker;
     * the 10th revision of the International Classification of Diseases (ICD-10) code;
     * medicines.
  3. Place index fingers on sensors that are on the case's backside and record 1-lead ECG of up to 3 minutes duration.
  Recorded parameters:
  * time parameters of the ECG intervals (RR, P, PR, QRS, QT, QTc);
  * abnormal rhythms;
    * heart rate variability;
    * additional function - blood pressure and blood sugar diary. All recorded and calculated parameters are passed to the server.

SUMMARY:
This interventional prospective multicenter nonrandomized clinical and epidemiological study is the first Russian study aimed at evaluating the effectiveness of a single-lead electrocardiography device (CardioQVARK) in screening for atrial fibrillation in primary health care.

DETAILED DESCRIPTION:
This is an interventional, prospective, multicenter, nonrandomized clinical and epidemiological study. We are planning to enroll 5,000 patients.

Three outpatient departments, 3 affiliates of a city clinical hospital and 6 rural health posts in Moscow region are equipped with 25 CardioQVARK electrocardiography (ECG) devises.

The study implies 9 stages:

1. Patient signs informed consent and consent to the processing of personal data than fills out a questionnaire in a mobile application (https://itunes.apple.com/ru/app/cardioqvark/id1320898122) and registers a 3-minute ECG with a single-lead CardioQVARK ECG device. If an episode of atrial fibrillation (AF) is not detected during a reception, but a patient describes symptoms of AF, we hand out the devices to such patients to take home with them.
2. All records that are registered at outpatient departments, affiliates, rural health posts and at home are sent to a server of "CardioQVARK" (Limited Liability Company). For data processing, an AF detecting algorithm is applied. If AF is detected, an ECG report is generated in PDF format.
3. Three independent cardiology experts receive ECG records and verify the performance of the algorithm. They decode and annotate ECG reports (PDF).
4. If the expert confirms that the algorithm detected an AF episode, the ECG report (PDF) is sent to an arrhythmologist for diagnosis. After that, the ECG record with confirmed diagnosis is passed to a physician at a health-care facility.
5. When the physician receives the report, he calls the patient to verify the diagnosis in a face-to-face consultation. That can be done by routine ECG, 24-, 48- or 72-hour ECG monitoring.
6. Anticoagulation therapy is revised or induced for all patients with diagnosed AF.
7. Six months after the enrollment, the patient is called for another face-to-face consultation with further peripheral venous blood sampling to assess anticoagulation therapy in terms of pharmacokinetics (assess compliance) and pharmacogenetics (assess the influence of genetic factors on anticoagulant effect of warfarin and new oral anticoagulants).
8. Estimating cost-effectiveness of using the single-lead CardioQVARK ECG device in screening for AF in primary health care.
9. Statistical processing of data and endpoints determination.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 18 to 96 years who have one or more of the following risk factors:

* hypertonic disease
* history of ischemic stroke or transient ischemic attacks
* type 1 and type 2 diabetes
* 1-3 degrees obesity
* heart failure or the presence of a clinic to reduce exercise tolerance associated with shortness of breath
* coronary heart disease or the presence of symptoms of chest pain, in the absence of an established diagnosis of coronary heart disease
* the presence of peripheral arterial atherosclerosis
* the presence of a clinic of interruptions in the work of the heart (bouts of rapid, irregular heartbeats, pauses in work of heart)

Non-inclusion criteria:

* Acute coronary syndrome
* Acute ischemic or hemorrhagic stroke
* Acute psychosis
* The presence of severe concomitant diseases with an expected life expectancy of less than 2 years

Exclusion Criteria:

Refusal of further participation in the study

Ages: 18 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Total number of AF cases newly diagnosed during the study period. | Through study completion, an average of 1 year
  Total number of AF cases newly diagnosed during the study period.
Number of patients who, for the first time ever, were assigned to anticoagulation therapy. | Through study completion, an average of 1 year
  Number of patients who, for the first time ever, were assigned to anticoagulation therapy.
Compliance to anticoagulation therapy for warfarin. | 6 months after administration of anticoagulants
  Assessed using data obtained from pharmacokinetic analysis. International normalised ratio (INR) - target range from 2 to 3.
Compliance to anticoagulation therapy for new oral anticoagulants. | 6 months after administration of anticoagulants
  Assessed using data obtained from pharmacokinetic analysis. Quantitative determination of the concentration of drugs in the blood (blood sampling three hours after taking the drug).
Cost-effectiveness of using the single-lead CardioQVARK ECG device in screening for AF in primary health care. | Through study completion, an average of 1 year
  Evaluated as incremental cost-effectiveness ratio of screening per quality adjusted life year gained, and per stroke avoided.

SECONDARY OUTCOMES:
Mean time to diagnosis. | Through study completion, an average of 1 year
  Mean time to diagnosis.
Number of patients with a CHA₂DS₂-VASc score (the CHA2DS2-VASc Score is the most commonly utilized method to predict thromboembolic risk in atrial fibrillation) of ≥ 1. | Through study completion, an average of 1 year
  Number of patients with a CHA₂DS₂-VASc score (the CHA2DS2-VASc Score is the most commonly utilized method to predict thromboembolic risk in atrial fibrillation) of ≥ 1.
Number of patients with a CHA₂DS₂-VASc score (the CHA2DS2-VASc Score is the most commonly utilized method to predict thromboembolic risk in atrial fibrillation) of ≥ 2. | Through study completion, an average of 1 year
  Number of patients with a CHA₂DS₂-VASc score (the CHA2DS2-VASc Score is the most commonly utilized method to predict thromboembolic risk in atrial fibrillation) of ≥ 2.
Incidence of ischemic stroke or transient ischemic attack after enrollment in the study. | Through study completion, an average of 1 year
  Defined as frequency of ischemic stroke or transient ischemic attack in patients with newly diagnosed AF and assigned anticoagulants.
Incidence of massive hemorrhage after enrollment in the study. | Through study completion, an average of 1 year
  Defined as frequency of massive hemorrhage in patients with newly diagnosed AF and assigned anticoagulants.
Incidence of hemorrhagic stroke after enrollment in the study. | Through study completion, an average of 1 year
  Defined as frequency of hemorrhagic stroke in patients with newly diagnosed AF and assigned anticoagulants.
Pharmacogenetic testing by polymorphic markers | 6 months after administration of anticoagulants
  * For warfarin - CYP2C9 (CYP2C9 * 2, CYP2C9 * 3), VKORC1 (1 marker), CYP4F2 (1 marker), GGCX (1 marker).
  * For new oral anticoagulants - rs2244613 of the gene CES1, rs1045642 (C3435T), rs1128503 (C1236T), rs2032582 (G2677T / А) of the gene ABCB1, rs2231142 (С421А, Q141K) of the gene ABCG2, rs776746 (A6986G * 399 CYP3 CYP3) CYP3A4.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Kopylov, Professor, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (12):
- Russia (12):
  - State Budgetary Healthcare Institution of Moscow Region "Mytishchi City Clinical Hospital", Mytishchi, Belyaninovo Village, Central Str., 41
  - State Budgetary Healthcare Institution of Moscow Region "Mytishchi City Clinical Hospital", Mytishchi, Boltino Village, Building 91
  - Clinic №2, State Budgetary Healthcare Institution of Moscow Region "Mytishchi City Clinical Hospital", Mytishchi, Microdistrict of the Village Pirogovskiy, Sovetskaya Str.
  - Branch of State Budgetary Healthcare Institution of Moscow Region "Mytishchi City Clinical Hospital", Mytishchi, Ostashkovo Village, Kashtanovaya Str., Possession 44.
  - State Budgetary Healthcare Institution of Moscow Region "Mytishchi City Clinical Hospital", Mytishchi, Pestovo Village, Berezovaya Alleya Str., 4, Room 15.
  - Branch office of State Budgetary Healthcare Institution of Moscow Region "Mytishchi City Clinical Hospital", Mytishchi, Povedniki Village, Lane Ovrazhny, Building 4.
  - State Budgetary Healthcare Institution of Moscow Region "Mytishchi City Clinical Hospital", Mytishchi, Troitskoye Village, Sel'skaya Str., Building 32.
  - Branch office of State Budgetary Healthcare Institution of Moscow Region "Mytishchi City Clinical Hospital", Mytishchi, Turpansionata Village, Turpansionata KVH, Sorokinskoe Highway
  - State Budgetary Healthcare Institution of Moscow Region "Mytishchi City Clinical Hospital", Mytishchi, Udino Village, Cvetochnaya Str., 3.
  - State Budgetary Healthcare Institution of Moscow Region "Mytishchi City Clinical Hospital", Mytishchi, Vitenevo Village, 58.
  - Clinic №1, State Budgetary Healthcare Institution of Moscow Region "Mytishchi City Clinical Hospital", Mytishchi
  - Clinic №4, State Budgetary Healthcare Institution of Moscow Region "Mytishchi City Clinical Hospital", Mytishchi

IPD SHARING:
Plan to Share IPD: No
The research sponsor is Sechenov University. Data disclosure is not permitted by the local ethics committee.
  For more information about the study, you need to contact the principal investigator.